CLINICAL TRIAL: NCT01776385
Title: Detection and Characterization of Circulating Tumor Cells in Patients With Malignant Pleural Mesothelioma: Towards a New Phase in the Understanding of the Natural History of This Cancer?
Brief Title: The ISET (Isolation by Size of Epithelial Tumor Cells) and the CellSearch Methods in Malignant Pleural Mesothelioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-AOI-08
Record Dates: First submitted 2012-03-23; First posted 2013-01-28 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-02

CONDITIONS: Pleural Neoplasms; Mesothelioma; Pneumothorax; Parathyroid Neoplasms; Benign Tumor of the Thyroid; Tumor of the Thyroid
Keywords: [C08.785.640]; (C08.528.778); [C19.642.713]; mesothelium
MeSH Terms: conditions — Pleural Neoplasms; Mesothelioma; Pneumothorax; Parathyroid Neoplasms; Thyroid Neoplasms | interventions — Blood Specimen Collection; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group patients (Experimental): Patients with Malignant Pleural Mesothelioma (all stages)
  Interventions: Other: Blood sampling
- Control group (Placebo Comparator): Patients with pneumothorax or of benign tumor of the thyroid
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Blood sampling — Biological: ISET and CellSearch Methods Sampling of blood - ISET and CellSearch Methods
  Arms: Group patients
Other: Control Group — Biological: ISET and CellSearch Methods Sampling of blood - ISET and CellSearch Methods
  Arms: Control group

SUMMARY:
Malignant pleural mesothelioma (MPM) has a growing incidence and in spite of early diagnostic, their outcome remains dismal. The evolution of MPM is often local with rare distant metastases. There is now a sizable body of evidence that metastases could develop from circulating tumor cells (CTC) spread in blood before or during surgery. Thus, sensitive and specific detection of CTC in blood is considered as a potentially relevant predictive biomarker for patients with carcinomas. In exchange, the prognostic value of CTC in MPM has not yet been evaluated.

Indeed, the main goal for preoperative detection of CTC is to identify patients with high risk of recurrence after surgery, in order to perform more adapted therapeutic strategy. Despite several studies reported about CTC detection, methodological aspects concerning sensitivity, specificity and reproducibility have prevented a clear appraisal of their clinical impact. Thus, the aim of our study is to evaluate the presence and the prognostic value of CTC in MPM by a double approach. In our setting, cytopathological analysis of circulating non hematological cells (CNHC), of epithelial origin, isolated according to their size (ISET, Isolation by Size of Epithelial Tumor cells) along with immunomagnetic selection, identification and enumeration of circulating epithelial cells in peripheral blood (CellSearch method) is considered a promising approach.

ELIGIBILITY:
Inclusion Criteria

For the patients:

* Age > 18 years
* Patient having been operated for a strong suspicion of a pleural malignant tumoral lesion corresponding to a primitive pleural mesothelioma
* Signed patient consent

For the control subjects:

* Age > 18 years
* unhurt of any malignant or mild tumoral pathology or patients that must benefit from a surgical procedure for a benign lesion in other organ than the pleura or a pulmonary non tumoral lesion
* Signed patient consent

Exclusion Criteria :

* Patient with histories of cancer or the other synchronous cancer
* Patient with additives treatments
* Patient according to treatments additives others than protocols codified (in particular, platinum navelbine or gemcitabine platinum) for stages II
* HIV, hepatitis B or C infections
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of presence / absence of CTC on the global survival | from Baseline in Systolic Blood Pressure at 6 months
  Value forecasts of the presence / absence of CTC on the global survival estimated by the estimation and the test of meaning at 0 of the immediate relative risk (fate ratio) in a model at proportional risk.

SECONDARY OUTCOMES:
Value forecasts of the number of CTC on the global survival estimated by the risk | from Baseline in Systolic Blood Pressure at 6 months
  Value forecasts of the number of CTC on the global survival estimated by the immediate relative risk Value forecasts of the presence / absence and the number of CTC on the survival without second offense(recurrence) or metastasis estimated by the immediate relative risk

CONTACTS AND LOCATIONS:
Overall Officials: ILIE Marius, PhD, Principal Investigator — LPCE- Hôpital de Pasteur - CHU de Nice
Locations (1):
- CHU de Nice - LPCE- Hôpital de Pasteur - 30 ave de la voie Romaine, Nice, Alpes-Maritimes, France